CLINICAL TRIAL: NCT05858827
Title: To Evaluate the Capability of an Endoscopic Ultrasonography Automatic Image Reporting System
Brief Title: To Evaluate the Capability of an EUS Automatic Image Reporting System
Status: Completed | Type: Observational
Sponsor: Renmin Hospital of Wuhan University (Other)
Responsible Party: Sponsor
Other Study IDs: EA-23-004
Record Dates: First submitted 2023-05-05; First posted 2023-05-15 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Endoscopic Ultrasonography; Artificial Intelligence
Keywords: Endoscopic Ultrasonography; Artificial Intelligence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, the EUS intelligent picture reporting system can automatically generate reports after reading videos of EUS examinations. This function can standardize the quality of endoscopic ultrasound image reporting and reduce the work burden of ultrasound endoscopists.

DETAILED DESCRIPTION:
A well-written report is the most important way of communication between clinicians, referring doctors and patients. Reports play a key role for quality improvement in digestive endoscopy, too. Unlike digestive endoscopy, the quality of reporting in endoscopic ultrasound (EUS) has not been thoroughly evaluated and a reference standard is lacking. According to the guidance statements regarding standard EUS reporting elements developed and reviewed at the Forum for Canadian Endoscopic Ultrasound 2019 Annual Meeting, appropriate photo documentation of all relevant lesions and anatomical landmarks should be included in EUS reports and stored for future reference. Systematic photo documentation in EUS is an indicator of procedure quality according to the ASGE. Systematic photo documentation can facilitate surveillance EUS evaluations. According to an international online survey, most endosonographers used a structured tree in the report describing either normal and abnormal findings (81%) or only abnormal findings (7%). Therefore, it is necessary to develop a standardized endoscopic ultrasound image report system.

The past decades have witnessed the remarkable progress of artificial intelligence (AI) in the medical field. Deep learning, a subset of AI, has shown great potential in elaborating image analysis. In the field of digestive endoscopy, deep learning has been widely studied, including identifying focal lesions, differentiating malignant and non-malignant lesions, and so on. However, rare study works on automatic photo documentation during endoscopic ultrasound.

Our previous work has successfully developed a deep learning EUS navigation system that can identify the standard stations of the pancreas and CBD in real time. In the present study, we further constructed an EUS automatic image reporting system (EUS-AIRS). The EUS-AIRS can automatically capture images of standard stations, lesions, and biopsy procedures, and label Types of lesions, thereby generating an image report with high completeness and quality during endoscopic ultrasonography.

We tested the performance of the EUS-AIRS by testing its performance on retrospective internal and external data, and we anticipate determining the utility of the EUS-AIRS in clinical practice by testing its performance in consecutive prospective patients.

ELIGIBILITY:
Inclusion Criteria:

1. patients aged 18 years or older;
2. patients with indications for endoscopic ultrasonography of the biliary pancreatic system and undergoing sedated EUS procedures;
3. ability to read, understand, and sign informed consent;

Exclusion Criteria:

1. patients with absolute contraindications to EUS examination;
2. history of previous gastric surgery;
3. pregnancy;
4. severe medical illness;
5. previous medical history of allergic reaction to anesthetics;
6. stricture or obstruction of the esophagus;
7. anatomical abnormalities of the upper gastrointestinal tract due to advanced neoplasia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population was patients undergoing endoscopic ultrasonography who met all inclusion criteria and did not meet all exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2023-05-10 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
completeness of capturing standard stations | 2 months
  The number of standard stations correctly captured by EUS-AIRS is divided by the number of all standard stations in the endoscopic ultrasound procedures

SECONDARY OUTCOMES:
accuracy of capturing standard stations | 2 months
  The number of standard station images correctly captured by EUS-AIRS is divided by the number of all standard station images captured by EUS-AIRS
completeness of capturing detected lesions | 2 months
  The number of correct lesions captured by EUS-AIRS was divided by the number of all lesions in the endoscopic ultrasound procedure
completeness of capturing biopsy procedures | 2 months
  The number of correct biopsy procedures captured by EUS-AIRS was divided by the number of all biopsy procedures in the endoscopic ultrasound procedure

CONTACTS AND LOCATIONS:
Overall Officials: Honggang Yu, Doctor, Principal Investigator — Renmin Hospital of Wuhan University
Locations (1):
- Renmin Hospital of Wuhan University, Wuhan, Hubei, China